CLINICAL TRIAL: NCT02209831
Title: An Open Label, Randomised, Crossover Study of the Bioavailability of Oral BIRB 796 BS Tablets (30 mg Single Dose) With and Without Administration of Oral Pantoprazole in Healthy Male Volunteers to Assess the Effect of Gastric pH on Absorption of BIRB 796 BS.
Brief Title: Bioavailability of Oral BIRB 796 BS Tablets With and Without Administration of Oral Pantoprazole in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1175.17
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Pantoprazole

ARMS (2):
- BIBR 796 BS + pantoprazole (Experimental)
  Interventions: Device: BIBR 796 BS; Drug: Pantoprazole
- BIBR 796 BS without pantoprazole (Active Comparator)
  Interventions: Device: BIBR 796 BS

INTERVENTIONS:
Device: BIBR 796 BS — single dose
Drug: Pantoprazole — 5 days
  Arms: BIBR 796 BS + pantoprazole

SUMMARY:
Study to assess the effect of gastric pH on the pharmacokinetics of BIRB 796 BS.

Safety and tolerability were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >=18 and <=55 years
* Laboratory examinations within a clinically defined reference range
* Helicobacter pylori negative
* Able to tolerate pH probe application
* Body mass index (BMI) >=18.5 and <=29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* Surgery of gastrointestinal tract (excluding appendectomy)
* History of orthostatic hypotension, fainting spells or blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator including study drugs
* History of vasculitis (past history of fever, malaise, myalgias, rash, etc.)
* Intake of drugs with a long half-life (> 24 hours) within 1 month or 10 half lives of that drug, whichever is longer, prior to administration of study drugs or during the trial
* Use of any drugs that might influence the results of the trial within 10 days prior to administration or during the trial
* Use of grapefruit or grapefruit juice, alcohol, green tea, methylxanthine-containing products or tobacco within 5 days of study drug administration
* Participation in another trial with an investigational drug within 1 month prior to administration or during the trial
* Smoker
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood or plasma donation (>400 ml) within 1 month prior to administration or during trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Following specific laboratory findings: aspartate aminotransferase, alanine transaminase, Gamma-glutamyl-transferase above the reference range
* Inability to comply with dietary regimen of study centre
* Inability to comply with investigator's instructions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2001-11; Primary Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve from time 0 mathematically extrapolated to time infinity (AUC0-inf.) | up to 36 hours after drug administration

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | up to 36 hours after drug administration
Area under the plasma concentration versus time curve over a given time interval (AUC0-t) | up to 36 hours after drug administration
Time to the maximum plasma concentration (tmax) | up to 36 hours after drug administration
Apparent oral clearance (CL/F) | up to 36 hours after drug administration
Apparent volume of distribution during the terminal elimination phase, divided by F (bioavailability factor) (Vz/F) | up to 36 hours after drug administration
Elimination half-life (t1/2) | up to 36 hours after drug administration
Mean residence time (MRT) | up to 36 hours after drug administration
Gastric pH measurements | up to 12 hours after drug administration
Number of patients with adverse events | up to 34 days
Assessment of tolerability | on the last 1 day of second treatment
  based on the ability of the subjects to take the medicine as well as occurence of adverse events and abnormal laboratory investigations

REFERENCES:
- See also: Related Info — http://clintriage.rdg@boehringer-ingelheim.com